CLINICAL TRIAL: NCT05836207
Title: The Cost-effectiveness of Contingency Management Compared to Standard Cognitive Behavioral Treatment for Treating Cannabis Use Disorder in Youth: A Randomized Controlled Trial
Brief Title: Rewards for Cannabis Abstinence-study
Acronym: RECAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parnassia Addiction Research Centre (Other)
Collaborators: Leiden University Medical Center (Other); Brijder Verslavingszorg (Unknown); Antes (Unknown); Novadic-Kentron (Unknown); Amsterdam University of Applied Sciences (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Trimbos (Unknown); Het Zwarte Gat (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10390012110082
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cannabis Use Disorder
Keywords: contingency management; cognitive behavioural therapy; CM; CBT; cost-effectiveness; youth; randomized controlled trial (RCT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abstinence-focused Contingency Management (CM) (Experimental): Youths receive 12 weeks of outpatient abstinence-focused CM consisting of providing incentives for cannabis abstinence, based on twice-weekly rapid test urinalysis.
  Interventions: Behavioral: Abstinence-focused Contingency Management (CM) - stand alone
- Cognitive Behavioural Therapy (CBT) (Active Comparator): Youths receive 12 weeks of outpatient usual care CBT consisting of once-weekly 60-minute sessions according to the standard CBT youth protocol by a trained psychologist.
  Interventions: Behavioral: Standard Outpatient Cognitive Behavioural Therapy (CBT)

INTERVENTIONS:
Behavioral: Abstinence-focused Contingency Management (CM) - stand alone — Outpatient abstinence-focused contingency management (CM) as stand-alone treatment (12 weeks). Monetary incentives (vouchers) are provided for cannabis abstinence, based on twice-weekly rapid test urinalysis and an escalating reward scheme with bonuses. Urine samples are collected at the treatment centre during 15-minute sessions by a trained CM-practitioner. For each cannabis-negative urine, patients receive a monetary voucher starting at €5 and escalating to max. €35 after eight consecutive weeks of cannabis abstinence, with an additional €10 bonus after two consecutive cannabis-negative urines. The voucher-value is reset to €5 after a cannabis-positive urine test. Total earnings can be max. €675 for 12 weeks of consecutive cannabis abstinence (average: €8 p/day). Youths sign an agreement stating that vouchers must be spent on recovery-oriented goals.
  Arms: Abstinence-focused Contingency Management (CM)
Behavioral: Standard Outpatient Cognitive Behavioural Therapy (CBT) — CBT is the usual care first line treatment for CUD in youth, in the Netherlands. CBT for CUD is focused on learning cognitive, emotional, motivational and behavioral skills to reduce or cease cannabis use, and generally consists of 12 once-weekly 60-minute sessions and 'homework' exercise assignments, provided by a psychologist.
  Youths receive 12 weeks of outpatient usual care CBT consisting of once-weekly 60-minute sessions according to the standard CBT youth protocol by a trained psychologist. CBT-youths receive the same cannabis urine-testing procedures as CM-youths, but test results will not be disclosed to treatment staff or patient, and no rewards will be given for cannabis abstinence.
  Arms: Cognitive Behavioural Therapy (CBT)

SUMMARY:
The goal of this clinical trial is to investigate the (cost-)effectiveness of contingency management (CM) compared with Cognitive Behavioural Therapy (CBT) for the treatment of cannabis use disorder (CUD) in youth (16-22 years).

The main questions it aims to answer are:

* What is the efficacy of 12 weeks outpatient CM versus CBT in youths with a CUD, in terms of cannabis abstinence during the intervention period?
* What is the long-term efficacy of CM versus CBT at 6- and 12-months follow-up (FU)?
* What is the cost-effectiveness of CM versus CBT at 12-months FU from a societal perspective?

Study hypotheses are:

1. CM will result in more cannabis-abstinent days than CBT during the intervention; 2. CM is more effective and cost-effective than CBT at 12 months follow-up.

Eligible patients (n=154) will be randomly assigned to either 12 weeks of outpatient CM or CBT. Assessments are conducted by trained research-assistants at baseline, after 6, 12, 26 and 52 weeks, and twice-weekly during treatment and consist of questionnaires, a computer task and collection of urine samples. Primary endpoint is the number of biochemically verified cannabis abstinent days in the 12-week treatment period. Key secondary endpoint: Treatment response: 50% or more reduction in cannabis use days in the past 4 weeks, compared with baseline.

The primary outcome will be modelled in the intention-to-treat population in a (negative binomial) regression analysis with treatment group as independent variable and stratification variables as covariates.

Cost-effectiveness and cost-utility analysis (CEA; CUA) will be performed from a societal perspective. CEA: Treatment response is the central clinical endpoint for calculations of incremental costs per responder. CUA: Incremental costs per QALY (based on EuroQoL).

ELIGIBILITY:
Inclusion Criteria:

* Youths (16-22 years) seeking treatment for a primary CUD
* Regular cannabis use (≥14 days) in past 4 weeks
* Intention to cease cannabis use during intervention
* Able and willing to attend the treatment center and submit urine samples under supervision twice-weekly
* Informed consent.

Exclusion Criteria:

* Health contra-indications (e.g., acute psychosis/suicidality)
* Insufficient Dutch language.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Cannabis-abstinent days (biochemically verified) | 12 weeks
  Number of biochemically verified cannabis-abstinent days during the 12-week intervention period

SECONDARY OUTCOMES:
long-term 'treatment response' | 52 weeks
  defined as 50% or more reduction in cannabis use days in the 4 weeks preceding week 12 (end-of-treatment), and week 26 and 52, compared with baseline.
Incremental costs per treatment responder | 52 weeks
  Incremental cost-effectiveness ratio (ICER) per treatment responder (see above) will be determined based on the incremental costs and effects of CM compared with CBT.
Incremental costs per QALY | 52 weeks
  Incremental costs per quality-adjusted life years (QALY) gains based on the The 5-level EQ-5D version (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Renske Spijkerman, PhD, Principal Investigator — PARC; Vincent Hendriks, Prof. dr., Study Director — PARC
Locations (5):
- Netherlands (5):
  - Jellinek, Stichting Arkin B.V., Amsterdam
  - IrisZorg, Arnhem
  - Antes Youz, Rotterdam
  - Brijder, The Hague
  - Novadic-Kentron, Vught

IPD SHARING:
Plan to Share IPD: Yes
First draft of datamanagement plan has been submitted to funding organisation.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: december 2028, 15 years